CLINICAL TRIAL: NCT06537648
Title: Decreasing Alzheimer's Risk Through oNline Choreographed Exercise - Down Syndrome
Acronym: DANCE-DS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: T32AG078114 (NIH)
Record Dates: First submitted 2024-07-18; First posted 2024-08-05 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Down Syndrome; Physical Inactivity
MeSH Terms: conditions — Down Syndrome; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decreasing Alzheimer's Risk Through oNline Choreographed Exercise - Down Syndrome (Experimental): Participants will be asked to play attend 35 minute, remotely delivered, group exercise classes using choreographed exercise twice a week for 12 weeks.
  Interventions: Behavioral: Decreasing Alzheimer's Risk Through oNline Choreographed Exercise - Down Syndrome Program

INTERVENTIONS:
Behavioral: Decreasing Alzheimer's Risk Through oNline Choreographed Exercise - Down Syndrome Program — Adults with Down syndrome will be asked to attend 35 minute, remotely delivered (Zoom®) group dance sessions twice weekly across 12 weeks. All sessions will be directed by an instructor experienced in leading 35 minute, group remote exercise sessions for individuals with intellectual disability as part of the ongoing exercise program for individuals with intellectual disability offered by the Division for Physical Activity and Weight Management.

SUMMARY:
The investigators are assessing acceptability, appropriateness, and feasibility of an remote choreographed exercise intervention using validated scales alongside qualitative data among young adults with Down Syndrome. Participants will take part in a 12-week exercise program with two 35-minute session per week delivered in a group setting. The aims of the project are to:

* Assess the feasibility of a 12 week remotely delivered group dance intervention.
* Assess changes in aerobic fitness and cognitive function in response to a 12 week remotely delivered group dance intervention.
* Assess the intensity and total energy expenditure of remotely delivered group dance sessions.

DETAILED DESCRIPTION:
The incidence of Alzheimer's disease for persons with Down syndrome exceeds 90%, and physical activity engagement has demonstrated potential to delay onset of Alzheimer's disease for this population. Adults with Down syndrome participate in less physical activity than their counterparts without disability, partially due to unique barriers preventing engagement in typical modalities of physical activity for this population. Dance, which is characterized by rhythmic physical movements offers the potential for social engagement, and stimulation of brain functions may offer a reasonable alternative to traditional physical activity modalities. However, empirical evidence to support the feasibility of a remotely delivered group dance intervention and evaluation of the intensity and energy expenditure achieved by a dance intervention for adults with Down syndrome are currently unavailable and will be the focus of the proposed pilot trial. Adults with Down will be asked to attend 35 minute remotely delivered (Zoom®) group dance sessions twice weekly across 12 weeks to assess the acceptability, appropriateness, and feasibility of the intervention, energy expenditure achieved during the exercise sessions, and evaluate change in aerobic fitness and cognitive function after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Down syndrome
* Sufficient functional ability to communicate through spoken language
* No plans to relocate outside the study area over the next 12 weeks
* Possession of a personal device that allows for connectivity to the internet and participate in 2x weekly group video calls
* Ability to participate in Moderate to vigorous physical activity

Exclusion Criteria:

* Serious medical risk (e.g., cancer, recent heart attack, stroke, pregnancy, angioplasty as determined by the research staff
* unwilling to participate in outcomes assessments
* uninterested

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Attendance | 12 weeks
  Attendance at each 35-minute online exercise classes will be collected. Attendance will be assessed as the number of sessions attended out of the total number of sessions available (24 sessions available).
Retention | 12 weeks
  Participant retention will be collected based on the number of participants who complete the 12 week intervention. A total of up to 20 participants will be enrolled into the study. Participants that complete the 12-week intervention will be considered retained. Any participant that discontinues participation prior to the end of the 12-week intervention will not be considered retained.
Adverse Events | 12 weeks
  Adverse events will be collected on a weekly basis.

SECONDARY OUTCOMES:
6-minute walk test | 12 weeks
  This test measures the distance that a participant can walk on a flat, hard surface in a period of 6 minutes. The research team will instruct them on how to prepare and conduct this test.
Episodic Memory | 12 weeks
  Episodic memory will be assessed before and after the intervention using the modified Cued Recall Test.
Energy Expenditure | 1 session
  Energy expenditure during a dance session (kilocalories per minute; Metabolic equivalents (METs) will be assessed by portable indirect calorimetry.
Exercise intensity | 12 weeks
  Exercise intensity will be assessed as an average of the percent of age-estimated maximal heart rate achieved during dance sessions assessed by a Fitbit®

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No